CLINICAL TRIAL: NCT01388205
Title: An Exploratory Randomized Controlled Trial of a Novel Family-Based Intervention to Increase Outdoor Time for the Prevention of Myopia and Increase Physical Activity Among Singapore Youth
Brief Title: Trial of a Novel Family-Based Intervention to Increase Outdoor Time and Fitness
Acronym: FIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Saw Seang Mei, Professor of Epidemiology, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FIT-NUS-10-520
Record Dates: First submitted 2011-06-30; First posted 2011-07-06 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Myopia; Obesity
Keywords: Myopia; Outdoor activity; Physical activity; Randomized Controlled Trial; Pedometer; Behavior modification; Obesity
MeSH Terms: conditions — Myopia; Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Family-based Intervention Arm (Experimental)
  Interventions: Behavioral: Family-based Outdoor program
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Family-based Outdoor program — 2 to 3 hour outdoor activities organized in conjunction with National Parks, Singapore
  Other Names: Outdoor intervention
  Arms: Family-based Intervention Arm

SUMMARY:
This study aims to implement a new family-based health behavior community program to increase time spent outdoors and physical activity among Singapore children aged 6 to 12 years in a 1-year randomized clinical trial. 300 children from 250 families will be randomly assigned to either a family-based intervention or no intervention. The family-based intervention comprises structured weekend outdoor activities organized by National Parks and incentives for children to wear a pedometer and increase their daily steps. Families who meet their monthly step and outdoor activity goals will receive a range of prizes and incentives. Both groups will receive brochures on the National Myopia Prevention Program and physical activity. The success of the intervention will be evaluated through light meters, 7-day outdoor diaries, questionnaires documenting outdoor time and myopia; as well as pedometer steps, walking tests, and body mass index. A community-based intervention will be developed to improve the health of Singapore children by increasing outdoor time and physical activity to prevent myopia and obesity.

DETAILED DESCRIPTION:
To develop, implement, and evaluate a novel incentive-based family intervention to increase time spent outdoors and physical activity among children aged 6 to 12 years in a 1-year randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Children between 6 and 12 years of age with no known health problems preventing them from staying outdoors or walking for physical activity will be included as long as they are Singapore citizens or permanent residents.
* Both myopic and non-myopic children will be included

Exclusion Criteria:

* Children with medical conditions such as Type 1 diabetes, severe asthma, cancer or mental illness will be excluded.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 285 (Actual)
Dates: Start 2011-04; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Physical fitness/Exercise capacity | Outcome measure will be assessed at baseline and 12 month follow-up visit
  Physical fitness/Exercise capacity assessed through 6-minutes walking test

SECONDARY OUTCOMES:
Outdoor time | Outcome measure will be assessed at baseline and 12 month follow-up visit
  Time spent outdoors assessed using the WHO Risk factor Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Saw Seang Mei, MBBS,PhD, Principal Investigator — National University of singapore, Department of Epidemiology & Public Health; Eric Andrew Finkelstein, PhD, Principal Investigator — Duke-NUS Graduate Medical School
Locations (1):
- National University of Singapore, Kent Ridge, Singapore

REFERENCES:
- [Derived] Finkelstein EA, Tan YT, Malhotra R, Lee CF, Goh SS, Saw SM. A cluster randomized controlled trial of an incentive-based outdoor physical activity program. J Pediatr. 2013 Jul;163(1):167-72.e1. doi: 10.1016/j.jpeds.2013.01.009. Epub 2013 Feb 14. PMID 23415616